CLINICAL TRIAL: NCT03404232
Title: The Use of the DTO Hybrid Dynamic Device: a Clinical Outcome- and Radiological-based Prospective Clinical Trial
Brief Title: Radiological and Clinical Efficacy of a Hybrid Spinal Implant ("Topping Off"): a Mono-center, Prospective Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Aachen (Other)
Responsible Party: Principal Investigator, Christian Herren, Principal Investigator, University Hospital, Aachen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKKuUKA001
Record Dates: First submitted 2018-01-05; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Spine Surgery

STUDY DESIGN:
Intervention Model Description: All patients requiring lumbar spinal surgery by the use of a hybrid spinal implant (DTO): (1) patients with their first surgical intervention at the lumbar spine, (2) patients with a previous surgical decompression but non-fusion procedure after LSS and (3) patients with medical history of PLIF-/TLIF-technique and later onset of symptomatic ASD within the superior adjacent segment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): patients with their first surgical intervention at the lumbar spine receive the Dynesys DTO device (Zimmer Spine, Inc.).
  Interventions: Device: Dynesys DTO device (Zimmer Spine, Inc.)
- Group 2 (Active Comparator): patients with a previous surgical decompression but non-fusion procedure after lumbar spinal stenosis surgery receive the Dynesys DTO device (Zimmer Spine, Inc.).
  Interventions: Device: Dynesys DTO device (Zimmer Spine, Inc.)
- Group 3 (Active Comparator): patients with the medical history of PLIF-/TLIF-technique and later onset of symptomatic ASD within the superior adjacent segment receive the Dynesys DTO device (Zimmer Spine, Inc.).
  Interventions: Device: Dynesys DTO device (Zimmer Spine, Inc.)

INTERVENTIONS:
Device: Dynesys DTO device (Zimmer Spine, Inc.) — All patients receive posterior hybrid instrumentation.

SUMMARY:
The study aim is to show the effectiveness of a hybrid system (DTO) regarding clinical outcome and radiological alteration in a single-center prospective setting.

DETAILED DESCRIPTION:
Posterior spondylodesis and monosegmental intervertebral cage plus flexible instrumentation of the superiorly adjacent segment (Dynesys DTO).

Planned follow-up visits up to 48 months with documentation of health-related outcome measurement instruments and radiological control of possible segment alteration and device-related complication.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Legal capacity
* Age ≥ 18 years
* Indication for monosegmental lumbar spine fusion (PLIF or "topping-off ") L2-S1 with osteochondrosis Modic grades I-III or spondylolisthesis Meyerding grades I-III.
* Radiologic signs of degeneration in the adjacent segment of the intended fusion without signs of instability

Exclusion Criteria:

* Motor deficit
* Cauda equina syndrome
* Previous surgical intervention of the lumbar spine
* Relevant peripheral neuropathy
* Acute denervation subsequent to a radiculopathy
* Scoliosis with Cobb angle greater than 25°
* Spondylolisthesis > Meyerding grade III
* Radiologic signs of degeneration in the adjacent segment of the intended fusion with signs of instability (for definition, see inclusion criteria)
* No radiologic signs of degeneration in the adjacent segment of the intended fusion (for definition, see inclusion criteria)
* Radiologic signs of degeneration in the adjacent segment of the intended fusion with >Fujiwara grade II or >Pfirrmann grade IV
* Signs of instability in any lumbar spine segment other than that undergoing fusion
* General contraindication for elective lumbar spine surgery
* Pathologic fracture
* Osteoporosis with pathologic fracture
* Active systemic infection
* Rheumatic disease
* Disease of bone metabolism (e.g. Paget's Disease)
* Bone metastasis
* Local infection focus lumbar spine
* Seizure disorder
* Chronic ischemia Fontaine classification IIb-IV
* Severe heart insufficiency (NYHA III-IV)
* Blood coagulation disorder or blood thinning therapy
* Cortisone intake more than one month in the last 12 months before randomization
* Simultaneous participation in another clinical trial in the 30 days before randomization
* Known allergy or intolerance to the implants
* Dependency on investigator
* Lack of familiarity with the German language
* Placement in an institution by governmental or juridical advice
* Absent legal capacity
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in the health-related outcome measurement instruments (ODI) | 24-48 months
Changes in the health-related outcome measurement instruments (COMI) | 24-48 months
Changes in the health-related outcome measurement instruments (SF-36) | 24-48 months
Radiological outcomes | 24-48 months
  Radiological changes within the adjacent segment

SECONDARY OUTCOMES:
Device complication (breakage, loosening, etc.) | 24 - 48 months
  Complication regarding the device
Patient-related complication | 24- 48 months
  general and surgical complication

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herren C, Sobottke R, Pishnamaz M, Scheyerer MJ, Bredow J, Westermann L, Berger EM, Oikonomidis S, Eysel P, Siewe J. The use of the DTO hybrid dynamic device: a clinical outcome- and radiological-based prospective clinical trial. BMC Musculoskelet Disord. 2018 Jun 21;19(1):199. doi: 10.1186/s12891-018-2103-x. PMID 30016956